CLINICAL TRIAL: NCT01819883
Title: Ectopic Lipid Deposition and Insulin Resistance in After Treatment of Acromegaly
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Assistant Physician in Medicine, Massachusetts General Hospital
Other Study IDs: 2012P002517
Record Dates: First submitted 2013-03-22; First posted 2013-03-28 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active Acromegaly: All study subjects with acromegaly will be studied twice - once during the active stage of their disease (pre-treatment) and a second time: 3 months after treatment of acromegaly. Controls will be studied at one time point.
- Healthy controls

SUMMARY:
This study investigates fat distribution in people with acromegaly. The investigator is also investigating the change of fat distribution before and after treatment of acromegaly. The investigator will compare the results of people with acromegaly to the results of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 75 yr (both groups)
* Study subjects with active acromegaly
* Healthy controls

Exclusion Criteria:

* Serum creatinine or alanine aminotransferase (ALT) > 2 times the upper limit of normal, metastatic cancer.
* Controls will be receiving no medications and have no chronic diseases, including cancer, hypertension or diabetes mellitus.
* Contraindications to MRI imaging (both groups) like those with certain metal implants, surgical clips or pacemakers.
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty-two study subjects will be studied: 1) patients with active acromegaly, and 2) healthy controls. Study subjects with acromegaly will be prescribed treatment for acromegaly by their healthcare providers, and this study will not interfere in anyway with clinical care and will not provide surgery, medications or other forms of clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy, matched controls completed a baseline visit only
Period: Overall Study
Arm/Group | Active Acromegaly | Healthy Controls
Started | 20 | 20
Completed | 16 | 20
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Acromegaly | Healthy Controls | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (16) | 47 (17) | 47 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 17 | 17 | 34
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Intrahepatic Lipids (Liver Fat) [Median (Inter-Quartile Range); unit: ratio] — Intrahepatic lipids are reported in lipid to water ratio units.
  ratio | 0.02 [0.01 to 0.04] | 0.06 [0.02 to 0.22] | 0.02 [0.01 to 0.09]
Intramyocellular Lipids (Muscle Fat) [Median (Inter-Quartile Range); unit: Arbitrary Units] | 8.2 [3.9 to 11.2] | 10.7 [6.4 to 14.1] | 9.5 [5.1 to 13.9]
Visceral Fat Area [Median (Inter-Quartile Range); unit: Cm^2] | 96 [62 to 188] | 140 [56 to 208] | 124 [59 to 205]
Thigh Muscle Cross-Sectional Area [Mean (Standard Deviation); unit: Cm^2] | 162 (38) | 158 (40) | 160 (39)
Fasting Insulin [Median (Inter-Quartile Range); unit: uU/mL] | 9 [7 to 17] | 6 [3 to 12] | 8 [4 to 14]
Insulin Area Under the Curve (AUC) [Median (Inter-Quartile Range); unit: uU/mLx120 min] | 6828 [5152 to 8196] | 3827 [1854 to 4580] | 4370 [2640 to 6350]
Insulin-like Growth Factor-1 (IGF-1) Blood Level [Median (Inter-Quartile Range); unit: ng/ml] | 787 [641 to 1099] | 174 [110 to 209] | 344 [174 to 809]

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Fat
Description: Change in intrahepatic fat after biochemical control of acromegaly
Time Frame: Baseline and 3-month follow-up visit
Population: 20 subjects with active acromegaly completed the baseline visit. 16 subjects completed the follow-up visit after biochemical control of acromegaly.
Measure: Median (Inter-Quartile Range); unit: Lipid/water ratio
Groups:
- Active Acromegaly: All study subjects with acromegaly will be studied twice - once during the active stage of their disease (pre-treatment) and a second time: approximately 3 months after treatment of acromegaly. Controls will be studied at one time point.
Arm/Group | Active Acromegaly
Number analyzed (Participants) | 16
Lipid/water ratio | 0.03 [0.01 to 0.30]

2. Primary Outcome: Change in Thigh Muscle Cross-sectional Area
Description: Change in thigh muscle cross-sectional area after biochemical control of acromegaly
Time Frame: Baseline and 3-month follow-up visit
Population: 20 subjects with active acromegaly completed a baseline visit. 16 subjects completed a follow-up visit after biochemical control of acromegaly had been achieved.
Measure: Mean (Standard Deviation); unit: Cm^2
Arm/Group | Active Acromegaly
Number analyzed (Participants) | 16
Cm^2 | 154 (45)

ADVERSE EVENTS:
Groups:
- Healthy Controls: Healthy, matched controls
Arm/Group | Active Acromegaly | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes